CLINICAL TRIAL: NCT04537195
Title: Effects on Anxiety and Depression of a Lay-led Transdiagnostic Self-management Program (ADSMP-C) for Patients Recently Treated for Cancer With Curative Intent: A Randomized Controlled Trial
Brief Title: Effects of a Lay-led Anxiety and Depression Self-management Program for Cancer Patients
Acronym: ADSMP-C
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: TrygFonden, Denmark (Industry); Komiteen for Sundhedsoplysning (Unknown); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 124941, TrygFonden; 2016-051-000001, ID 1174 (Other: Aarhus University, Denmark)
Record Dates: First submitted 2020-08-27; First posted 2020-09-03 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Neoplasms; Anxiety; Self Efficacy; Psychological Distress; Cancer; Distress, Emotional; Depression; Group, Peer
Keywords: Intervention; RCT
MeSH Terms: conditions — Neoplasms; Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blinded at 7-month follow-up when administering the Hamilton rating scales (secondary outcomes). Participants will be instructed not to disclose their group allocation until the interview is completed
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Experimental): ADSMP-C
  Interventions: Behavioral: ADSMP-C
- Control Group (No Intervention): Wait-list control group

INTERVENTIONS:
Behavioral: ADSMP-C — A transdiagnostic, lay-led, group-based self-management program consisting of seven 2 ½ hour weekly sessions focusing on increasing patient self-efficacy in symptom management of anxiety and depression in cancer (ADSMP-C)
  Arms: Intervention Group

SUMMARY:
The investigators aim to evaluate a peer-to-peer patient self-management program targeting symptoms of anxiety and depression in a randomized trial. A total of 234 cancer patients recently having completed primary treatment with curative intent in central Region Denmark will be included. The intervention is a lay-led, group-based transdiagnostic patient education program consisting of seven 2 ½ hour weekly sessions focusing on increasing patient self-efficacy in symptom management of anxiety and depression. The intervention is highly structured and manualized.

DETAILED DESCRIPTION:
Recent evidence suggest that transdiagnostic interventions may be just as effective as traditional diagnosis specific interventions when treating symptoms of depression and anxiety. Brief lay-led transdiagnostic self-management interventions may therefore offer an efficient alternative to traditional symptom specific interventions (e.g. CBT) when targeting symptoms of depression and anxiety in cancer.

The present study aim to evaluate The Anxiety and Depression Symptom Management Program (ADSMP) in a cancer setting (ADSMP-C). The ADSMP is a Danish adaptation of The Stanford University Chronic Disease Self-Management Program (CDSMP) and is developed by the Danish Health Information Committee (In Danish: Komiteen for Sundhedsoplysning in collaboration with The Expert Patient Program Community Interest Company (EPPCIC), the English Health Service (NHS) and Stanford University.

The ADSMP-C is a lay-led, group-based transdiagnostic patient education program consisting of seven 2 ½ hour weekly sessions focusing on increasing patient self-efficacy in symptom management of anxiety and depression concluded with a networking session. The intervention is highly structured and manualized. Sub-group analyses on participants with a history of cancer in a larger trial of ADSMP conducted by members of the study group on behalf of the Danish National Board of Health showed promising results. However, a larger study is needed to establish sound scientific evidence on the effectiveness of the program in a cancer setting.

A total 234 cancer patients recently having completed primary treatment with curative intent in central Region Denmark will be randomized (2:1) to ADSMP-C or a control arm respectively. As a part of the recruitment procedure patients will be screened with The "Distress-Thermometer" at the departments of oncology at the two largest hospitals in Central Region, Denmark following primary treatment or at a follow-up (< 1yrs. after primary treatment).

Participants completes online questionnaires (REDCap) at baseline (pre-randomization), at post-intervention, and at three (primary follow-up) and six months post-intervention, including the Beck's Depression Inventory (BDI-II) and Spielbergers State-Trait Anxiety Inventory (STAI-state) (primary outcomes). In addition, all participants will be interviewed at 7 month post-intervention. Outcome assessors, blind to group allocation, will perform observer-based Hamilton A6 and D6 short-form ratings at the interview (secondary outcomes).

Data will be evaluated by mixed-effects regression analyses (intention-to-treat).

The current study will be the first to evaluate the efficacy of ADSMP in a cancer setting.

ELIGIBILITY:
Inclusion Criteria:

* Treated in Central Region Denmark
* Recently completed (< 1 yr.) primary treatment for cancer with curative intent
* BDI-II score >=14 and/or STAI-state score >=40

Exclusion Criteria:

* Not sufficient Danish language skills to fill Questionnaires and participate in a group based intervention
* Psychosis
* Aggressive behavior
* Imminent suicidal risk

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2020-03-06 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Change in Depressive Symptoms | Baseline and 3 months post-intervention
  Beck Depression Inventory (BDI-II)
Change in Anxiety Symptoms | Baseline and 3 months post-intervention
  Spielberger State-Trait Inventory (STAI). State subscale.

SECONDARY OUTCOMES:
Change in Anxiety Symptoms | Baseline and 6 months post-intervention
  Spielberger State-Trait Inventory (STAI). State subscale.
Change in Depressive Symptoms | Baseline and 6 months post-intervention
  Beck Depression Inventory (BDI-II)
Change in Anxiety (observer-rated) | Baseline and 7 months post-intervention
  Hamilton Anxiety Rating Scale (HAM-A6)
Change in Depression (observer-rated) | Baseline and 7 months post-intervention
  Hamilton Depression Rating Scale (HAM-D6)
Change in Fear of cancer recurrence | Baseline and 3 months post-intervention
  Concerns About Recurrence Questionaire (CARQ-4)
Change in Self-efficacy - Personal control | Baseline and 3 months post-intervention
  The Revised Illness Perception Questionnaire (IPQ-R). Personal Control subscale.
Change in Self-efficacy - Social support | Baseline, and 3 months post-intervention
  Obtain Help from Community, Family, Friends Scale (SECD-Ssup)

CONTACTS AND LOCATIONS:
Overall Officials: Soren Christensen, MSc., Principal Investigator — Dep. Psychology, Aarhus University, Denmark
Locations (2):
- Denmark (2):
  - Dep. Oncology, Aarhus University Hospital, Aarhus
  - Dep. Oncology, Regional Hospital West Jutland, Herning

IPD SHARING:
Plan to Share IPD: No
At the present the policy of Aarhus University does not allow the sharing of data according to GDPR rules. However this policy may be subject to change